CLINICAL TRIAL: NCT00073164
Title: A Study of the Safety and Efficacy of Depakote ER Plus an Atypical Antipsychotic Vs. an Atypical Antipsychotic Alone in the Treatment of Schizophrenia
Brief Title: Depakote ER Plus an Atypical Antipsychotic Vs. an Atypical Antipsychotic Alone in the Treatment of Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M02-547
Record Dates: First submitted 2003-11-17; First posted 2003-11-18 (Estimated); Last update posted 2006-08-04 (Estimated); Status verified 2006-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine; Risperidone

INTERVENTIONS:
Drug: Divalproex Sodium Extended-Release Tablets
Drug: Olanzapine
Drug: Risperidone

SUMMARY:
The purpose of this study is to assess the 14-day and 12-week safety and efficacy of Depakote ER used in combination with either olanzapine or risperidone versus antipsychotic monotherapy with olanzapine or risperidone for the treatment of schizophrenia.

ELIGIBILITY:
KEY INCLUSION CRITERIA:

* Acute exacerbation of schizophrenia as defined by: subject recently hospitalized or is in the process of being admitted to a hospital or an acute care inpatient psychiatric treatment facility; and has a PANNS Total score of 70 or greater at the time of screening and at randomization based on a 1-7 point scale; and has a score on any two of the four items from psychosis cluster of the BPRS (extracted from the PANSS) that correspond to the positive symptoms (hallucinatory behavior, unusual thought content, conceptual disorganization and suspiciousness) totaling 8 or greater; and has a total of 6 or greater on one of the following two pairs of items from the BPRS (extracted from the PANSS): hostility and uncooperativeness or excitement and tension.
* Current DSM-IV-TR diagnosis of schizophrenia as confirmed by the SCID
* Positive response to antipsychotics in the previous 2 years

KEY EXCLUSION CRITERIA:

* Current diagnosis of schizoaffective disorder, drug-induced psychosis, manic episode or major depressive episode.
* At the time of screening, has been hospitalized for more than 14 days for the current episode
* Has ever taken clozapine
* Has had more than 3 psychiatric hospitalizations in the previous 6 months or has had more than 8 weeks of psychiatric hospitalization in the previous 12 months
* Has serious violent, homicidal, suicidal ideation
* Has received depot medications fluphenazine decanoate and/or haloperidol decanoate within 2 or 4 weeks prior to randomization respectively
* Urine toxicology screen is positive for phencyclidine (PCP), opiates, cocaine or amphetamines
* History of alcohol or substance dependence within the past month
* Has taken any valproate product for a psychiatric indication within the previous 30 days
* Has received an investigational drug within the last 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2003-07

PRIMARY OUTCOMES:
The psychiatric rating scale battery will include the PANSS, the CGI Scale, and the CDSS. The NOSIE, Overall Treatment Evaluation, Burden Questionnaire, and Quality of Life Scale.

SECONDARY OUTCOMES:
The movement rating scale battery will include the Simpson-Angus Scale (SAS), the Barnes Akathisia Scale (BAS), and the Abnormal Involuntary Movement Scale (AIMS).

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information 800-633-9110, Study Director — Abbott
Locations (35):
- United States (35):
  - Birmingham, Alabama
  - Tuscaloosa, Alabama
  - Anaheim, California
  - Cerritos, California
  - Chula Vista, California
  - Garden Grove, California
  - Glendale, California
  - Los Angeles, California
  - San Diego, California
  - Denver, Colorado
  - Gainsville, Florida
  - Melbourne, Florida
  - North Miami, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Indianapolis, Indiana
  - South Bend, Indiana
  - Shreveport, Louisiana
  - Rockville, Maryland
  - Jackson, Mississippi
  - Clementon, New Jersey
  - Kenilworth, New Jersey
  - Holliswood, New York
  - New York, New York
  - Butner, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Austin, Texas
  - Irving, Texas
  - San Antonio, Texas
  - Falls Church, Virginia